CLINICAL TRIAL: NCT04416269
Title: Use of Oral Antidiabetic Agents in Hospitalized Patients With Diabetes
Brief Title: Oral Anti Diabetic Agents in the Hospital
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Maya Fayfman, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00117027; 1K23DK124647-01 (NIH)
Record Dates: First submitted 2020-06-02; First posted 2020-06-04 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus
Keywords: Hyperglycemia; Insulin therapy; Oral therapy; Basal bolus therapy; Mean daily blood glucose; Hospitalization
MeSH Terms: conditions — Diabetes Mellitus; Hyperglycemia | interventions — Metformin; Sulfonylurea Compounds; Pioglitazone; Insulin Glargine; Insulin Detemir; Insulin Lispro; Insulin Aspart; Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Oral Anti-diabetes Drugs (OADs) alone (Experimental): OADs will be continued at same outpatient dosage unless contraindicated
  Interventions: Drug: Oral Anti-diabetes Drugs alone; Drug: Supplemental insulin; Device: Continuous glucose monitoring (CGM)
- Basal bolus insulin (Active Comparator): Basal insulin with glargine or detemir and rapid-acting insulin (lispro/aspart) will be used as per the hospital formulary. OADs and non-insulin injectable antidiabetic medication will be discontinued on admission.
  Interventions: Drug: Basal bolus insulin; Drug: Supplemental insulin; Device: Continuous glucose monitoring (CGM)

INTERVENTIONS:
Drug: Oral Anti-diabetes Drugs alone — OADs will be continued at same outpatient dosage unless contraindicated. Participants will be switched to the preferred drug within the category of medication they take at home. Dose adjustment for OADs will be based on clinical/laboratory status. The OAD will be held if the participant is placed on strict nil per os (NPO) and is unable to take oral medications after enrollment.
  Other Names: metformin; sulfonylureas; pioglitazone; dipeptidyl peptidase-4 (DPP-4) inhibitors; sodium-glucose co-transporter 2 (SGLT2) inhibitors
  Arms: Oral Anti-diabetes Drugs (OADs) alone
Drug: Basal bolus insulin — Basal insulin with glargine or detemir will be used as per the hospital formulary.
  Other Names: glargine; detemir
  Arms: Basal bolus insulin
Drug: Supplemental insulin — Supplemental (correction) lispro or aspart insulin following the supplemental/sliding scale standard of care protocol for BG >140 mg/dl.
  Other Names: Humalog; Novolog
Device: Continuous glucose monitoring (CGM) — A subset of participants (50 per study arm) will be randomized to take part in an optional study where a CGM device will be placed for the duration of the study. CGM reports will be reviewed at the end of the study to assess parameters of glycemic control and hypoglycemia, and not used for insulin dose adjustment.
  The Dexcom CGM is a small sensor that inserts just under the skin to continuously monitor glucose levels. Results are transmitted to the wearer's smartphone every five minutes.
  Other Names: Dexcom

SUMMARY:
This randomized controlled clinical trial will assess whether continuation of home oral antidiabetic agents during hospitalization can be used as a safe and effective alternative to insulin therapy in the management of diabetes in the hospital. The primary outcome of the study is to determine differences in glycemic control as measured by mean daily blood glucose concentration between oral antidiabetic medications and basal bolus therapy in hospitalized patients with type 2 diabetes (T2D).

DETAILED DESCRIPTION:
Hyperglycemia in the hospital is common and has been associated with increased hospital complications, length of stay, and mortality. Improving glycemic control has been shown to improve length of stay, multi-organ failure, systemic infections, as well as short- and long-term mortality. Clinical guidelines from professional organizations recommend the use of subcutaneous (SQ) insulin as the preferred therapy for glycemic control in general medical and surgical patients with T2D. This approach, however, is labor intensive requiring multiple daily insulin injections, costly, and associated with significant risk of iatrogenic hypoglycemia

Over 75% of patients with T2D are treated with oral antidiabetic drugs (OADs) but due to the lack of safety and efficacy data from randomized controlled trials, clinical guidelines recommend stopping OADs during hospitalization. The current clinical guidelines have raised concerns with the use of OADs including risk of hypoglycemia with sulfonylureas, fluid retention and worsening of heart failure with thiazolidinediones, and risk of metformin-associated lactic acidosis in patients with severe renal impairment. However, several observational studies have reported that the use of OADs results in similar glycemic control without increased risk of complications compared to insulin regimens. A recent observational study that included 17,325 hospitalized patients with T2D, found that patients treated with OADs had similar glycemic control without differences in complications and no increase in rates of hypoglycemia compared to those treated with insulin.

This study will assess whether continuation of home oral antidiabetic agents during hospitalization can be used as a safe and effective alternative to insulin therapy in the management of diabetes in hospital patients with T2D. For a subset of participants (50 patients per group), a CGM devise will be placed for the duration of the study to assess parameters of glycemic control and hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, age 18-80 years admitted to a general medicine and surgery services
* Known history of T2D receiving OADs either as monotherapy or in combination therapy
* Admission BG < 250 mg/dl or randomization BG <250 mg/dl and not receiving basal insulin
* Patients receiving OADs in combination with GLP-1 receptor agonists (GLP-1RA) who have HbA1c <7.5% within the past three months
* HbA1c <10%

Exclusion Criteria:

* No known history of diabetes
* Laboratory evidence of diabetic ketoacidosis
* Subjects with a history of type 1 diabetes (suggested by BMI < 25 requiring insulin therapy or with a history of diabetic ketoacidosis, or ketonuria)
* Meeting any exclusion criteria based on specific contraindications to their home oral therapy
* Acute critical illness or cardiac surgery expected to require admission to a critical care unit
* Gastrointestinal obstruction, adynamic ileus, or expected to require gastrointestinal suction
* Medical or surgical patients expected to be kept NPO for >24-48 hours after admission or after completion of surgical procedure
* Impaired renal function (eGFR <30 ml/min)
* Current treatment with oral or injectable corticosteroid
* Mental condition rendering the subject unable to understand the nature and scope of the study
* Female subjects who are pregnant or breastfeeding at time of enrollment in the study
* New or recent onset (within two weeks) of coronavirus disease 2019 (COVID-19) infection at the time of admission

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2020-08-07 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Mean daily BG concentration | During hospital stay (up to 10 days)
  Mean daily BG concentration will be compared between OADs and basal bolus therapy in hospitalized patients with T2D.

SECONDARY OUTCOMES:
Number of mild hypoglycemic events | During hospital stay (up to 10 days)
  Mild hypoglycemic events are defined as BG <70 mg/dl. Hypoglycemic events are assessed by point of care (POC) testing and continues glucose monitoring (CGM).
Number of clinically significant hypoglycemic events | During hospital stay (up to 10 days)
  Clinically significant hypoglycemic events are defined as BG <54 mg/dl. Hypoglycemic events are assessed by POC testing and CGM.
Number of severe hypoglycemic severe (<40 mg/dl) events | During hospital stay (up to 10 days)
  Severe hypoglycemic events are defined as BG <40 mg/dl. Hypoglycemic events are assessed by POC testing and CGM.
Percent of BG within target range without hypoglycemia | During hospital stay (up to 10 days)
  The percentage of BG values within the target range of 70-180 mg/dl and without hypoglycemia will be compared between study arms.
Number of episodes of hyperglycemia after the first day of treatment | During hospital stay (up to 10 days)
  The number of episodes of hyperglycemia (BG > 280 mg/dl) after the first day of treatment will be compared between study arms.
Daily dose of insulin | During hospital stay (up to 10 days)
  The total daily dose of insulin will be compared between study arms.
Number of patients using oral antidiabetic drugs (OADs) during hospitalization | During hospital stay (up to 10 days)
  The number of participants using OADs during hospitalization use will be recorded.
OAD dose used during hospitalization | During hospital stay (up to 10 days)
  Dosage of OADs used during hospitalization will be recorded.
Number of patients on OADs requiring insulin rescue therapy | During hospital stay (up to 10 days)
  The number of patients on OADs requiring insulin rescue therapy will be recorded
Number of episodes of treatment failure | During hospital stay (up to 10 days)
  Treatment failure is defined as mean daily BG > 240 mg/dl or 3 consecutive BG > 240 mg/dl.
Glycemic variability in participants receiving CGM monitoring | During hospital stay (up to 10 days)
  Glycemic variability will be measured using the coefficient of variation
Time above BG target range (>180 mg/dl) in participants receiving CGM monitoring | During hospital stay (up to 10 days)
  The percentage of time above BG target range (>180 mg/dl) will be assessed in participants receiving CGM monitoring.
Time in BG target range (70-180 mg/dl) in participants receiving CGM monitoring | During hospital stay (up to 10 days)
  The percentage of time in the BG target range (70-180 mg/dl) will be assessed in participants receiving CGM monitoring.
Time below BG target range (BG <70 mg/dl) in participants receiving CGM monitoring | During hospital stay (up to 10 days)
  The percentage of time below BG target range (BG <70 mg/dl) will be assessed in participants receiving CGM monitoring.
Number of hospital complications | During hospital stay (up to 10 days)
  Hospital complications is assessed as a composite variable including infectious, renal, pulmonary, neurologic, cardiovascular complications, and mortality.
In-hospital mortality | During hospital stay (up to 10 days)
  In-hospital mortality will be recorded will be compared between study arms.
Number of individual hospital complications | Up to 40 days (hospital stay plus 30 days after discharge)
  Number of individual hospital complications will be compared between study arms. The specific complications assessed for this outcome include acute respiratory failure, acute renal failure (incremental rise in creatinine by 0.5 mg/dL from baseline), infection during hospitalization not felt to be present on admission (including wound infection, urinary tract infection, bacteremia), myocardial infarction, cardiac arrhythmia, congestive heart failure, and cardiac arrest.
Hospital costs | During hospital stay (up to 10 days)
  Total hospital costs will be compared between study arms.
Length of hospital stay | During hospital stay (up to 10 days)
  Length of hospital stay, in days, will be compared between study arms.
Costs for diabetes specific therapies | During hospital stay (up to 10 days)
  Costs for diabetes specific therapies (including insulin, oral agents, and cost of injection administration) will be compared between study arms.
Number of hospital re-admissions | within 30 days of hospital discharge
  Number of hospital re-admissions within 30 days of hospital discharge will be compared between study arms.
Number of emergency room visits | within 30 days of hospital discharge
  Number of emergency room visits within 30 days of hospital discharge will be compared between study arms.
Number of participants requiring ICU care | During hospital stay (up to 10 days)
  The number of participants transferred to the ICU will be compared between study arms.
Nursing antihyperglycemic drug preference survey | Day of hospital discharge (up to 10 days)
  The nurse who provided the most care for the participant during hospitalization completed a 7-item survey assessing antihyperglycemic drug preference. Nurses indicate if they agree or disagree with statements related to patient outcomes, workload requirements of insulin therapy, and perceived usefulness and safety of OADs. A summary score is not calculated for this qualitative survey.
Patient antihyperglycemic drug preference survey | Day of hospital discharge (up to 10 days)
  Participants will complete a 2 to 5-item survey assessing preferences of antihyperglycemic medications while hospitalized. Participants indicate if they agree or disagree with statements about OAD and insulin use during hospital stays, timely administration of insulin, and concerns about low blood sugar. A summary score is not calculated for this qualitative survey.

CONTACTS AND LOCATIONS:
Overall Officials: Maya Fayfman, MD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Grady Memorial Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be available for sharing.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Individual participant data will be made available for sharing beginning 3 months and ending 5 years following article publication.
Access Criteria: Individual participant data will be made available for sharing to researchers who provide a methodologically sound proposal. The proposal should be directed to maya.fayfman@emory.edu. To gain access, data requestors will need to sign a data access agreement.